CLINICAL TRIAL: NCT00897286
Title: Molecular and Histopathologic Characterization of Atypical Teratoid Rhabdoid Tumors, Choroid Plexus Carcinomas, Ependymomas, Medulloblastoma HGNET, CNS Embryonal Tumors and Gliomas of the Pediatric CNS
Brief Title: Study of Stored Tumor Samples in Young Patients With Brain Tumors
Status: Terminated | Type: Observational
Why Stopped: New Protocol that replaces the current study
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NBTP01
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood atypical teratoid/rhabdoid tumor; childhood choroid plexus tumor; childhood medulloblastoma; recurrent childhood medulloblastoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood ependymoma; recurrent childhood supratentorial primitive neuroectodermal tumor; untreated childhood supratentorial primitive neuroectodermal tumor; gliomas
MeSH Terms: conditions — Central Nervous System Neoplasms; Rhabdoid Tumor; Choroid Plexus Neoplasms; Medulloblastoma; Familial ependymoma; Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh frozen, fresh and/or cryopreserved, fixed and cultured tumor cells collected prospectively from a clinically well characterized patient cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor/Tissue Sample: Tumor material collected prospectively from a clinically well characterized patient cohort

SUMMARY:
This laboratory study is looking at stored tumor samples in young patients with brain tumors. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
The overall objective of this non-therapeutic protocol is to develop and molecularly characterize patient-derived orthotopic xenografts (PDOXs), organoids and in vitro models derived from medulloblastomas, High Grade Neuroepithelial Tumors (HGNET), CNS embryonal tumors, Atypical Teratoid Rhabdoid Tumors (ATRTs), Choroid Plexus Carcinomas (CPCs), ependymomas, and gliomas. The investigators will characterize the genome-wide mutation, expression and epigenetic signatures of these models and compare them with the primary tumors from which they were derived, thus creating a well-characterized and invaluable resource for research on these rare and deadly pediatric brain tumors. This will also provide important insights into intratumoral heterogeneity, and molecular abnormalities that may influence the selective pressures driving evolution, and tumor growth as in PDOXs, organoids or in vitro cultures and define the relationship between these abnormalities and tumor histologic and clinical characteristics. This objective will be achieved by applying state-of-the-art DNA, RNA and epigenome analysis tools to the study of fresh frozen and/or cryopreserved, fixed and cultured tumor cells, PDOXs and organoids. The establishment of patient-derived orthotopic xenografts, organoids and cell cultures from each tumor sample will also allow for in vitro and in vivo analysis of tumor cell growth, signaling and therapeutic response.

ELIGIBILITY:
Inclusion Criteria

* Tumor may be primary, progressive or recurrent CNS tumor including brain and/or spine. All tumor types will be included with a focus on medulloblastoma, HGNET, CNS embryonal tumors, gliomas, ependymoma, CPC and ATRT tumors. Low grade gliomas are currently very challenging to culture and implant but if techniques mature these will also be included. Although rare, patients with ATRT may present with a primary renal and CNS tumor. In these instances samples will be collected from both the kidney and CNS tumor for analysis if available.
* Tumor may be collected at surgery prior to histologic confirmation
* Age less than 40 years at the time of initial diagnosis.
* Enrollment in the current version of the institution's banking protocol

Exclusion Criteria

* Diagnosis of tumor outside the central nervous system.
* Age greater than or equal to 40 years at the time of diagnosis

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will all brain tumor types will be included with a focus on medulloblastoma, HGNET, CNS embryonal tumors, gliomas, ependymoma, CPC and ATRT tumors. All studies will be conducted using tumor material collected prospectively from a clinically well characterized patient cohort.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2004-11-30 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Relationship between molecular abnormalities and tumor histologic and clinical characteristics | 20 Years

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols